CLINICAL TRIAL: NCT06835881
Title: Exploratory Study on the Value of Advanced Respiratory Monitoring Data During Mechanical Ventilation in Patients With Acute Respiratory Distress Syndrome (ARDS) in Terms of (1) Estimating the Risk of Ventilator Induced Lung Injury (VILI) and (2) the Relationship Between Aeration Benefit and Gas Exchange
Brief Title: Prevention of Lung Injury Induced by Mechanical Ventilation in Acute Respiratory Distress Syndrome ARDS Patients
Acronym: PULMODEL
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241678
Record Dates: First submitted 2025-01-09; First posted 2025-02-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Adult Respiratory Distress Syndrome
Keywords: Ventilator optimization; Ventilator induced lung injury; Digital twin; Smart data
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Given the huge volume of mechanically ventilated patients at risk of ARDS, optimizing hematosis by limiting pulmonary and systemic aggression associated with artificial ventilation techniques is a key objective if we are to further improve the prognosis of ARDS.

With a view to improving cardiopulmonary monitoring in ARDS, modeling using digital twins individualized by nature should ultimately enrich the diagnostic approach by simplifying the technical set-up. Advances in modeling in terms of speed, rendering and results could be applied to personalized monitoring to find the right artificial ventilation setting for the right patient, at the right time.

DETAILED DESCRIPTION:
During mechanical ventilation (MV) of patients with acute respiratory distress syndrome (ARDS), the application of the most protective ventilatory strategy possible, based on the reduction of volotrauma and the personalized prescription of a positive end-expiratory pressure (PEEP) regime, is the guarantee of clinical benefit, demonstrated in terms of tidal volume in particular (reduced mortality and number of days without mechanical ventilation).

When a benefit for patients with ARDS is found in clinical trials, it is mainly related to a reduction in the damage caused by mechanical ventilation.

Through technological progress mechanical ventilation optimization is guided by advanced monitoring, including measurement of transpulmonary pressure (TPP or LP) and/or functional imaging data (e.g. Electro-impedance Tomography, EIT).

All these monitoring systems are now incorporated in the new generation of ventilators.

* Transpulmonary pressure (TPP); By estimating trans-pulmonary pressure, investigators can assess pulmonary stress and, without doubt, better interpret critical alveolar opening pressure.
* Continuous measurement of lung pressures and volumes (end-expiratory lung volume, EELV, as a substitute for functional respiratory capacity (FRC)) can also be obtained using more recent techniques based on the study of exhaled CO2 kinetics (volumetric capnography and dynamic capnometry).
* Electro-Impedance Tomography (EIT) ; Electrical impedance tomography (PulmoVista 500 ® , Drager, Germany; or integrated into the respirator, ELISA800VIT® , Lowenstein, Germany) provides totally non-invasive, cross-sectional visualization of part of pulmonary aeration, both dynamically and regionally.

This observational study on clinical physiological data is based on the reuse of pseudonymized recorded data in 1st-line care during sequential diagnostic maneuvers based on calibrated variations in PEEP and tidal volume and obtained by advanced respiratory monitoring in the acute phase of ARDS (esophageal manometry and/or EIT) and in accordance with the most recent recommendations.

No specific research procedures are planned for this study. This study will be conducted exclusively on the basis of personal data collected as part of the usual monitoring of a participant with ARDS undergoing advanced respiratory care. The analysis focuses on data recorded during recruitment maneuvers performed as part of care for this type of patient in the ICU.

Participants are informed individually, and their non-objection to the re-use of their data for research purposes is recorded in the file. Where applicable, information is given to the trusted support person/relative/parent if the participant is unable to express his/her wishes and does not object to the re-use of his/her data for research purposes. An information note is given to the patient or the trusted support person/relative/parent

Monitoring data is currently available in the Clinical Research Unit of our Intensive Care Departments, thanks to a data extraction system based on PHILIPS IntelliVue® or Mindray Benevision® monitoring solutions. It should be noted that the Data Warehouse Connect software solution enables all these data to be collected with fine sampling (2 ms for tracings, 1s for digital data), considerably extending the capabilities in terms of data analysis and exploitation. The extraction system is temporally coupled to patient events and medication (doses) administered, thanks to an IntelliSpace Critical Care and Anesthesia (ICCAA) information system that is operational in the ICU.

These data are downloaded onto a secure server with restricted access, then loaded into a database (SQL) for future processing of the pseudonymized data.

The data will be collected as part of routine care and is integrated in compliance with the RGPD.

Demographic data will be collected using the intensive care record (ORBIS or equivalent / computerized patient record).

Aim of the study Does the analysis of advanced monitoring data provide characteristic measured parameters that could help prevent or even reduce ventilator-induced lesions? Can these data be integrated into a model to build a digital twin for practical, simplified monitoring of ventilatory function?

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years requiring intensive care hospitalization for moderate-to-severe ARDS defined by a PaO2/FiO2 ratio < 200 mmHg and benefiting from respiratory monitoring including esophageal pressure (EPP) and EIT.
* Patient having been individually informed and not objecting to the re-use of his/her data for research purposes or, where applicable, trusted support person / close relative / parent of patient unable to express his/her wishes.

Exclusion Criteria:

* Patient, or where applicable, trusted support person / close relative / parent of patient unable to express his/her wishes, opposed to the re-use of his/her data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants or populations are selected based on predefined criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Describe and a posteriori analyze the recorded data and establish a relationship between the biomechanical characteristics of the data ("air" compartment, stress and strain) and the risk of mechanical ventilation-induced lesions (MVIL) in ARDS patients. | Acquisition and recording of monitoring data up to 5 days of intensive care in the acute phase of ARDS.
  - PEEP levels (cmH2O)

SECONDARY OUTCOMES:
Describe and a posteriori analyze the data recorded and establish a relationship between aeration gain and gas exchange. | Acquisition and recording of monitoring data up to 5 days of intensive care in the acute phase of ARDS
  Ventilation/pulmonary perfusion (in %) obtained with the Electro-Impedance Tomography (EIT) data
Use part of the collected data to customize a continuously calibrated integrative biomechanical model of the cardiopulmonary system to create a digital twin of the patient. | Acquisition and recording of monitoring data up to 5 days of intensive care in the acute phase of ARDS.
  - Transpulmonary pressure (TPP) (in cmH2O)
Stratify physiological data according to the main phenotypes determining respiratory mechanics, or endotypes of interest, for a personalized approach to ventilator settings (active and passive phases). | Acquisition and recording of monitoring data up to 5 days of intensive care in the acute phase of ARDS.
  - Pulmonary stress (mL/cmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice VALLEE, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France

IPD SHARING:
Plan to Share IPD: No